CLINICAL TRIAL: NCT05401903
Title: Measurement of Heart Rate Variability During Chiropractic Maintenance Care: Relationship Between Chiropractic Care and Autonomic Nervous System Regulation
Brief Title: Relationship Between Chiropractic Care and Autonomic Nervous System Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeast College of Health Sciences (Other)
Responsible Party: Principal Investigator, Jeanmarie R. Burke, PhD, Dean of Research and Faculty, Northeast College of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-02
Record Dates: First submitted 2022-05-29; First posted 2022-06-02 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Chiropractic Maintenance Care and Heart Rate Variability
Keywords: chiropractic; autonomic nervous system; healthy subjects

STUDY DESIGN:
Intervention Model Description: Pragmatic feasibility trial comparing the effects of chiropractic maintenance care versus a control group, no chiropractic care, on heart rate variability in healthy male adults.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chiropractic Maintenance Care (Experimental): The intervention group will receive weekly chiropractic care, in the form of high-velocity, low amplitude (HVLA) chiropractic adjustments delivered to restricted vertebrae of the cervical, thoracic and lumbar spinal segments. The intervention duration is 8 weeks. Subjects in the intervention group who do not attend at least four (4) scheduled chiropractic visits will be withdrawn from the study.
  Interventions: Other: Chiropractic Maintenance Care
- Control (No Intervention): The control group will not receive any chiropractic care during study protocol.

INTERVENTIONS:
Other: Chiropractic Maintenance Care — Subjects will receive high-velocity, low amplitude (HVLA) chiropractic manipulations to areas of defined restriction in the upper cervical spine, thoracic spine, lumbar spine, and pelvis. The clinician will use motion palpation to determine spinal segments with joint restrictions. Subjects will schedule weekly chiropractic visits.
  The clinician will not use passive care modalities. The exclusions of passive modalities include heat and cold therapies, electric stimulation, massage, acupuncture, and cupping therapies. Subjects will be encouraged to maintain normal exercise activity levels throughout the study. The clinician will provide instructions on homecare exercises as needed to promote range of motion of spinal segments between chiropractic visits. A single clinician will deliver the HVLA chiropractic manipulations to ensure consistency of chiropractic care throughout the study.
  Arms: Chiropractic Maintenance Care

SUMMARY:
The objective for this study is to explore the utility of biometric devices to measure changes in heart rate variability (HRV) during chiropractic maintenance care. The study will use WHOOP wearable technology to measure HRV. Chiropractic maintenance care refers to regular visits to manage recurrent musculoskeletal pain and dysfunction [1]. Beyond managing pain and dysfunction, regular chiropractic visits may also promote improvements in homeostatic regulation of internal physiological conditions, but the evidence-based is lacking for these effects [2]. The hypothesis of this study is that chiropractic maintenance care may lead to an increase in HRV as compared to a control group that do not receive chiropractic care.

1. Eklund A, Jensen I, Lohela-Karlsson M, Hagberg J, Leboeuf-Yde C, Kongsted A, et al. The Nordic maintenance care program: Effectiveness of chiropractic maintenance care versus symptom-guided treatment for recurrent and persistent low back pain-a pragmatic randomized controlled trial. PLoS One. 2018;13:e0203029.
2. Kovanur Sampath K, Mani R, Cotter JD, Tumilty S. Measureable changes in the neuro-endocrinal mechanism following spinal manipulation. Med Hypotheses. 2015;85:819-24.

DETAILED DESCRIPTION:
The study design is a pragmatic feasibility trial comparing the effects of chiropractic maintenance care versus a control group, no chiropractic care, on heart rate variability (HRV) in healthy male adults. The subjects in both groups will be healthy controls as the purpose of the study is to determine beneficial effects, if any, of chiropractic maintenance care on physiological function as opposed to pain management. The theoretical framework suggests a potential role of chiropractic maintenance care in the prevention of segmental dysfunction in the spine and cascading neuro-endocrine responses to biomechanical stress of the spinal segments, hypomobility [1, 2].

Chiropractic maintenance care will be for a duration of 8 weeks with subjects scheduled for one visit per week. Control subjects will be asked to refrain from chiropractic care for 8 weeks. All subjects will be asked to maintain the current status of their lifestyle behaviors for the duration of the study period, e.g. do not change diet or exercise training schedules. Using the WHOOP wearable technology to record daily HRV, the primary outcome is the weekly average of HRV. There will be a baseline week of HRV recordings prior to starting the intervention phase of the study. An increase in HRV of at least 6.5% from baseline to 8 weeks without a concomitant change in the control group will provide preliminary insights on chiropractic maintenance care and regulation of autonomic nervous system functions. As this is a feasibility study to explore the utility of biometric devices to measure changes in HRV during chiropractic maintenance care, sample size is limited to 20 subjects.

The 20 subjects will be healthy male adults from 18 to 40 years old. Given the small sample size. females are being excluded to avoid any confounding effects of menstrual cycle on the measurement of HRV. The summary of the evidence to date indicates medium to large effects in fluctuations of HRV across the menstrual cycle [3]. The study design will include simple randomization of subjects into chiropractic maintenance care or control group. The intervention group will receive weekly chiropractic care, in the form of high velocity, low amplitude (HVLA) chiropractic adjustments delivered to restricted vertebrae of the cervical, thoracic and lumbar spinal segments. Motion palpation of the spine will be used to identify restricted vertebrae of the cervical, thoracic and lumbar spinal segments. Subjects in the intervention group who do not attend at least four (4) scheduled chiropractic visits will be withdrawn from the study. Subjects in the control group who receive more than two (2) chiropractic treatments (visits) will be withdrawn from the study. Subjects in either group who receive more than two (2) other complementary and alternative (CAM) therapies (visits) will be withdrawn from the study.

1. Kovanur Sampath K, Mani R, Cotter JD, Tumilty S. Measureable changes in the neuro-endocrinal mechanism following spinal manipulation. Med Hypotheses. 2015;85:819-24.
2. Sampath KK, Botnmark E, Mani R, Cotter JD, Katare R, Munasinghe PE, et al. Neuroendocrine response following a thoracic spinal manipulation in healthy men. J Orthop Sports Phys Ther. 2017;47:617-27.
3. Schmalenberger KM, Eisenlohr-Moul TA, Würth L, Schneider E, Thayer JF, Ditzen B, et al. A systematic review and meta-analysis of within-person changes in cardiac vagal activity across the menstrual cycle: Implications for female health and future studies. J Clin Med. 2019;8.

ELIGIBILITY:
Inclusion Criteria:

1. Males, Minimum age of 18 years and Maximum age of 40 years
2. Subjects with access to a smart phone for use with the WHOOP app to allow for data tracking throughout the study.
3. Subjects are willing to be randomized to either the experimental group, maintenance chiropractic care, or control group, no chiropractic care.
4. Subjects are willing to not participate in other complementary and alternative medicine (CAM) therapies during the study period.

Exclusion Criteria:

1. Females.
2. Any diagnosed medical condition.
3. Any prescription medication use.
4. Have a pacemaker or other internal electronic device.
5. Any acute musculoskeletal (MSK) injuries involving the back and upper and lower extremities (e.g., neck, mid-back, lower back, shoulder, elbow, wrist, hand, hip, knee, ankle, foot etc.).
6. Any chronic MSK injuries involving the back and upper and lower extremities, (e.g., neck, mid-back, lower back, shoulder, elbow, wrist, hand, hip, knee, ankle, foot etc.).
7. Any contraindications to receive high velocity-low amplitude (HVLA) chiropractic manipulations.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | Nine Weeks
  Using the WHOOP wearable technology, daily Heart Rate Variability calculated during sleep will be recorded and averaged by week

OTHER OUTCOMES:
Strain | Nine Weeks
  Using the WHOOP, daytime Strain will be recorded daily and averaged by week
Heart Rate | Nine Weeks
  Using the WHOOP wearable technology, heart rate during sleep, upon waking, during activities of daily living and during exercise will be extracted from the daily heart rate profile. Average heart rate and maximum heart rate will be recorded during each defined interval on a daily basis and averaged by week.
Calories Burned | Nine weeks
  Using the WHOOP wearable technology, daytime calories will be recorded and averaged by week
Sleep | Nine weeks
  Using the WHOOP wearable technology, daily hours of sleep will be recorded and averaged by week
Respiratory Rate | Nine weeks
  Using the WHOOP wearable technology, daily respiratory rate (median) during sleep will be recorded and averaged by week.
Blood Oxygen Level | Nine weeks
  Using the WHOOP wearable technology, daily blood oxygen levels during sleep will be recorded and averaged by week.
Lifestyle Behaviors | Nine weeks
  Using the WHOOP Journal, self-reported changes in nutrition, activities of daily living, exercise training schedules, and the use of complementary and alternative therapies. Completed daily. Qualitative review to detect any major changes in lifestyle behaviors during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanmarie Burke, PhD, Study Director — Northeast College of Health Sciences
Locations (1):
- Jeanmarie R Burke, Seneca Falls, New York, United States